CLINICAL TRIAL: NCT03270527
Title: Reading Imperial Surrey Saturated Fat Cholesterol Intervention (RISSCI) Study. RISSCI-1 Blood Cholesterol Response Study
Brief Title: RISSCI-1 Blood Cholesterol Response Study
Acronym: RISSCI-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: University of Reading (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, Bruce A. Griffin, Professor, University of Surrey
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: RN0307A
Record Dates: First submitted 2017-08-10; First posted 2017-09-01 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Lipids; Lipid Metabolism; Healthy
Keywords: Dietary fat modification; Lipids; LDL cholesterol; Dietary fatty acids; Saturated fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High SFA diet to low SFA diet (Experimental): Participants will undergo, sequentially, a high SFA diet (Diet 1) followed by a low SFA diet (Diet 2) for 4 weeks each. Study visits will occur before and after each dietary intervention period. To comply with current UK dietary recommendations, Diets 1 and 2 will both contain ~35% energy from total fat. These diets will be consumed within the homes of free-living participants, by the substitution of ~40g of habitual fat, with either SFA-rich or mono/poly-unsaturated fatty acid-rich (MUFA/PUFA) cooking oils, spreads and snack foods, while maintaining their habitual diet (consistent intake of protein and carbohydrates, including dietary fibre). This will be achieved using a dietary exchange model developed and peer-reviewed for a previous dietary intervention study ('DIVAS') at the University of Reading, U.K.
  Interventions: Other: High SFA diet (Diet 1); Other: Low SFA diet (Diet 2)

INTERVENTIONS:
Other: High SFA diet (Diet 1) — 'Diet 1' will contain ~18% of its total energy as SFA .
Other: Low SFA diet (Diet 2) — 'Diet 2' will contain ~10% of its total energy as SFA. The SFA-replacement fats will be mixture of PUFA/MUFA.

SUMMARY:
Raised blood cholesterol (also referred to as blood LDL-cholesterol) is a major risk factor for developing heart disease. Dietary saturated fat is recognised as the main dietary component responsible for raising blood LDL-cholesterol, and reducing its intake has been the mainstay of dietary guidelines for the prevention of heart disease for over 30 years. However, there is very little evidence for a direct link between the intake of saturated fat and risk of dying from heart disease. One explanation for this, is that the link between saturated fat intake and heart disease is not a direct one, but relies heavily on the ability of saturated fat to raise blood LDL-cholesterol levels. This LDL cholesterol-raising effect of saturated fat is complex, and highly variable between individuals because of differences in the metabolism of dietary fat and cholesterol between people. The main aim of this study is to measure the amount of variation in blood LDL-cholesterol in healthy volunteers at the Universities of Surrey and Reading in response to lowering the amount of saturated fat in the diet to the level recommended by the government for the prevention of heart disease. This collaborative project between the Universities of Reading, Surrey and Imperial ('RISSCI-1' Blood Cholesterol Response Study') will permit identification of two subgroups of men who show either a high or low LDL-cholesterol response to a reduction in dietary saturated intake. These two groups of participants will be provided with an opportunity to participate in a similar follow-up study ('RISSCI-2') that will also take place at the University of Surrey and Reading. In this follow-up study, the participants will be asked to repeat a similar study protocol as for RISSCI-1, but undergo more detailed measurements to investigate the metabolic and genetic origins of how saturated fat is metabolised in the body and influences blood LDL-cholesterol (LDL-C).

DETAILED DESCRIPTION:
The LDL cholesterol-raising effect of saturated fatty acids (SFA) is complex, and highly variable between individuals because of differences in the metabolism of dietary fat and blood cholesterol between people. While these differences in metabolism make it difficult to study how dietary SFA influences LDL-cholesterol in large numbers of people, they can be measured in the laboratory and used as biological markers to distinguish between people who respond well from those who will respond less well to moderate-fat diets, which are lower in SFA.

The main aim of this study is to measure the amount of variation in blood LDL-cholesterol in healthy male volunteers in response to the replacement of SFA with unsaturated fats, and to select LDL-C responders from non-responders for a subsequent metabolic study ('RISSC-2'). Estimate of statistical power and sample size for 'RISSCI-1': A decrease of 0.16 mmol/L (SD 0.54) in our primary outcome of fasting plasma LDL-C between the high- and low-SFA diets, as observed in a previous randomly controlled trial, will require a sample size of 92 participants, at 80% power and 5% significance level. An estimated attrition rate of 15% will increase this sample size to 106 participants. To recruit this sample of participants, we anticipate having to screen 150 volunteers (75 at each site).

Specific objectives:

1. Undertake a dietary intervention study to examine the effects of two, 4 week diets that differ in their composition of fatty acids. The first diet ('Diet 1') will contain ~18% of its total energy as saturated fatty acids (SFA), while the second diet ('Diet 2') will contain ~10% of its total energy as SFA. Blood, urine and stool samples taken at the beginning (week 0) and end of Diet 1 (week 4), and end of Diet 2 (week 8), will be analysed to measure blood LDL-cholesterol and other relevant blood, urine and faecal metabolites. The white blood cell buffy coat will also be isolated from the blood samples collected at the baseline visit to enable genotyping of relevant genes involved in the absorption and metabolism of dietary fat.
2. To examine the data for evidence of associations between the changes in blood LDL- cholesterol, and the physical and biochemical characteristics of the participants as possible determinants of the variation in serum cholesterol response. This will include measurement of a common genetic polymorphism in APOLIPOPROTEIN E, as an established determinant of variation in blood cholesterol in response to dietary SFA.
3. To identify two subgroups of individuals whose blood LDL-cholesterol either responds ('Responders') or show little or no response ('Non-responders') on changing from Diet 1 to Diet 2, for participation in the follow-up study ('RISSCI-2'), which will be conducted at the Universities of Surrey, Reading and Imperial College London. In this follow-up study, the participants will be asked to repeat a similar study protocol as for RISSCI-1, and undergo more detailed measurements to determine how saturated fat is metabolised in the body.

Hypothesis:

In accordance with the variation in blood LDL-cholesterol response, that many studies have reported previously following substitution of dietary saturated with unsaturated fats, the investigators hypothesise that consuming Diet 1 (a high saturated fat diet) for 4 weeks followed by diet 2 (a low saturated fat/high unsaturated fat diet) for a further 4 weeks, will: 1) produce a variable distribution of responses in LDL-cholesterol that will enable the study of associations between the participants' baseline characteristics as possible determinants of the observed variation in blood LDL-cholesterol response, and 2) identify two distinct subgroups of individuals who either respond or show little or no response in their blood LDL- cholesterol. These distinct groups will be defined by the top and bottom ~10% of change in the concentration of blood LDL-cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 19-32 kg/m2
* Fasting serum total cholesterol < 7.5 mmol/l and triacylglycerol < 2.3 mmol/l

Exclusion Criteria:

* Smokers
* Medical history of myocardial ischemia or stroke in the past 12 months;
* Diabetes (defined as fasting glucose > 7.0 mmol/l) or other endocrine disorders; kidney, liver, pancreas or gastrointestinal disorders
* Hypertension (blood pressure > 140/90 mmHg),
* Cancer
* Medication for hyperlipidaemia (e.g. statins), hypertension, inflammation or prescribed antibiotics within the last three months
* Drinking in excess of 14 units of alcohol per week,
* Anaemia (<130 g/L haemoglobin), or planning on a weight-reducing regime
* Taking any dietary supplements known to influence lipids/gut microbiota (eg. plant stanols, fish oil, phytochemicals, natural laxatives, probiotics and prebiotics)
* Any other unusual medical history or diet and lifestyle habits or practices that would preclude volunteers from participating in a dietary intervention and metabolic study.

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in fasting total cholesterol (consisting of LDL-cholesterol and HDL) concentrations | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)

SECONDARY OUTCOMES:
Fasting triacylglycerol | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
HDL immune functions | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
HDL anti-inflammatory and anti-oxidant (PON-1) properties | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
HDL capacity to promote cholesterol efflux (ex-vivo) | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
Fasting insulin, glucose | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
Adhesion molecules, markers of vascular function | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
Inflammatory markers & adipokines | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
LDL-R gene expression | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
Other relevant genes involved in the absorption and metabolism of dietary fat | Baseline
  Polymorphic genes with potential influence on the serum LDL response to dietary saturated fat, e.g.: ATP-binding cassette proteins (cholesterol efflux proteins) ABCG5 (e.g. C1950G) ABCG8 (e.g. D19H, C1895T), functional polymorphisms in the farnesoid X receptor (FXR) and bile acid transporters (e.g. solute carrier organics anion 1B1). Fatty acid desaturases (FADS1 and FADS2). The patatin-like phospholipase domain-containing protein (PNPLA3) (e.g. rs738409 C/G), eNOS. Lipid/cholesterol homeostasis: serum apolipoprotein genes: APOE (ε2,ε3,ε4 e.g. rs429358 and rs7412), APOA-I (e.g. -75G/A), APOA4 (e.g. 360-2), APOA5 (e.g. -113/T&gt:c), APOCIII, APOB (e.g. -516C/T). Lipase genes: (e.g. LPL, HL, MGLL). Lipoprotein receptor genes (e.g. pvu11 in the LDL receptor), lipid transfer proteins (e.g. CETP e.g Taq1B, MTP), and other polymorphic genes related to the absorption and metabolism of dietary fat and regulation of lipid/cholesterol homeostasis.
Metabolomic analysis for the determination of the low molecular weight metabolite profiles in the biological fluids | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
  Analyses conducted by Imperial College London
Changes in faecal bacterial population | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
Weight | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
  BMI will also be calculated (kg/ height in m^2)
Fat mass | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
Fat free mass | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
Waist circumference | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
Hip circumference | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
Blood pressure | Baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
Fasting vascular stiffness | baseline, 4 weeks (after diet 1), 8 weeks (after diet 2)
  Measured via pulse wave assessment using the Mobil-O-graph device.

OTHER OUTCOMES:
Genotyping for apolipoprotein E to determine the impact of this genotype on changes in the primary and secondary outcome measurements in response to dietary fat intake | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Griffin, PhD, Principal Investigator — University of Surrey; Julie Lovegrove, PhD, Principal Investigator — University of Reading
Locations (2):
- United Kingdom (2):
  - Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire
  - Department of Nutritional Sciences, University of Surrey, Guildford, Surrey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vafeiadou K, Weech M, Altowaijri H, Todd S, Yaqoob P, Jackson KG, Lovegrove JA. Replacement of saturated with unsaturated fats had no impact on vascular function but beneficial effects on lipid biomarkers, E-selectin, and blood pressure: results from the randomized, controlled Dietary Intervention and VAScular function (DIVAS) study. Am J Clin Nutr. 2015 Jul;102(1):40-8. doi: 10.3945/ajcn.114.097089. Epub 2015 May 27. PMID 26016869
- [Derived] Koutsos A, Griffin BA, Antoni R, Ozen E, Sellem L, Wong G, Ayyad H, Fielding BA, Robertson MD, Swann J, Jackson KG, Lovegrove JA. Variation of LDL cholesterol in response to the replacement of saturated with unsaturated fatty acids: a nonrandomized, sequential dietary intervention; the Reading, Imperial, Surrey, Saturated fat Cholesterol Intervention ("RISSCI"-1) study. Am J Clin Nutr. 2024 Oct;120(4):854-863. doi: 10.1016/j.ajcnut.2024.07.032. Epub 2024 Aug 5. PMID 39111551
- [Derived] Sellem L, Antoni R, Koutsos A, Ozen E, Wong G, Ayyad H, Weech M, Schulze MB, Wernitz A, Fielding BA, Robertson MD, Jackson KG, Griffin BA, Lovegrove JA. Impact of a food-based dietary fat exchange model for replacing dietary saturated with unsaturated fatty acids in healthy men on plasma phospholipids fatty acid profiles and dietary patterns. Eur J Nutr. 2022 Oct;61(7):3669-3684. doi: 10.1007/s00394-022-02910-2. Epub 2022 Jun 6. PMID 35668120

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT03270527/Prot_SAP_000.pdf